CLINICAL TRIAL: NCT04293198
Title: PROOF: Evaluating the Performance of the KODEX-EPD CRyOballoon Occlusion Feature in Patients With Atrial Fibrillation
Brief Title: Evaluating the Performance of the KODEX-EPD CRyOballoon Occlusion Feature in Patients With Atrial Fibrillation
Acronym: PROOF
Status: Completed | Type: Observational
Sponsor: EPD Solutions, A Philips Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-KODEX-0019
Record Dates: First submitted 2020-02-20; First posted 2020-03-03 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Atrium; Fibrillation; Ablation
Keywords: Atrial Fibrillation; AF; Cryoballoon; Ablation; KODEX-EPD
MeSH Terms: conditions — Atrial Fibrillation | interventions — Fluoroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- control arm: Cryoballoon PVI procedure where the freeze was initiated based on the occlusion assessed using fluoroscopy
  Interventions: Device: Fluoroscopy with contrast dye
- Kodex arm: Cryoballoon PVI where the freeze was initiated based on the outcome of the KODEX occlusion Viewer
  Interventions: Device: KODEX-EPD System

INTERVENTIONS:
Device: KODEX-EPD System — The KODEX - EPD system is an open platform that uses any validated EP catheter to create real-time 3D images of the human heart. The KODEX occlusion viewer provides an indication of the occlusion status of the PV during cryoballoon PVI procedure
  Other Names: KODEX Occlusion Viewer
  Groups: Kodex arm
Device: Fluoroscopy with contrast dye — Fluoroscopy with contrast dye is used to determine occlusion status during cryoballoon PVI procedures
  Groups: control arm

SUMMARY:
Prospective, multi-center, non-randomized, open label, double arm study to assess the performance of the KODEX-EPD PV occlusion viewer. This study includes patients with atrial fibrillation who are scheduled to undergo a cryo balloon ablation procedure for their atrial fibrillation.

DETAILED DESCRIPTION:
The study is designed to evaluate the performance of the KODEX-EPD occlusion viewer using a standardized workflow in a blinded setting in a homogenous patient group. Furthermore, in an effort to minimize therapy, a direct comparison between the success of the freeze when initiating therapy based on the occlusion viewer vs the assessment of occlusion assessed with fluoroscopy will be evaluated. The study design indicates a post-market interventional clinical investigation to evaluate the endpoints of the study. No follow-up is foreseen ensuring a minimal burden to the subjects participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be aged >18 years.
2. Subject must have signed a written Informed Consent form to participate in the study, prior to any study related procedures.
3. Subject must be willing to comply with the protocol requirements.
4. Subject receives a de novo ablation procedure for treatment of atrial fibrillation.

Exclusion Criteria:

1. Pregnant women.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Arrhythmia patients scheduled to undergo a cryo balloon ablation procedure for their atrium fibrillation. Both male and female subjects who meet all eligibility criteria and give written informed consent will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the KODEX-EPD Occlsuion Viewer | up to approximately 6 months
  The primary effectiveness endpoint is the accuracy, sensitivity, specificity and positive and negative predictive values of the KODEX-EPD PV occlusion feature as compared to conventional angiographic method of fluoroscopy with contrast dye that will be used to guide the procedure.
Freeze success of the KODEX-EPD Occlusion Viewer | up to approximately 6 months
  The success of the freeze when freeze is initiated based on the assessment of the KODEX-EPD PV occlusion feature as compared to the success of the freeze when freeze is initiated based on the assessment with fluoroscopy and contrast dye.

CONTACTS AND LOCATIONS:
Locations (2):
- John Hopkins University, Baltimore, Maryland, United States
- UZ Brussel, Brussels, Belgium

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/98/NCT04293198/Prot_SAP_000.pdf